CLINICAL TRIAL: NCT00070447
Title: Phase II Study of Rituximab (NSC 687451) + CHOP Followed by 90Y-Ibritumomab Tiuxetan (NSC 710085) in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Rituximab, Prednisone, Cyclophosphamide, Doxorubicin, Vincristine, and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Previously Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000334470; ECOG-E1499
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2004-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab and yttrium Y 90 ibritumomab tiuxetan, can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy, such as prednisone, cyclophosphamide, doxorubicin, and vincristine, use different ways to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab and combination chemotherapy together with yttrium Y 90 ibritumomab tiuxetan works in treating patients with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the time to treatment failure in patients with previously untreated mantle cell lymphoma treated with rituximab and CHOP chemotherapy comprising prednisone, cyclophosphamide, doxorubicin, and vincristine followed by yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8; yttrium Y 90 Zevalin®).
* Determine the response rate in patients at the completion of rituximab and CHOP and the incremental response rate after IDEC-Y2B8.
* Determine the toxicity of this regimen in these patients.
* Correlate serum rituximab levels with response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* CHOP chemotherapy and rituximab: Patients receive cyclophosphamide IV, doxorubicin IV, vincristine IV, and rituximab IV on day 1 and oral prednisone on days 1-5 (R + CHOP). Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who have responding or stable disease proceed to radioimmunotherapy.

* Radioimmunotherapy: Within 4-7 weeks after the completion of R + CHOP chemotherapy, patients receive rituximab IV and an imaging dose of indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients then undergo whole body gamma imaging scans during the first day (2-24 hours) and the second or third day (48-72 hours) after injection. In the absence of altered biodistribution, patients receive rituximab IV followed by yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8; yttrium Y 90 Zevalin®) IV over 10 minutes on day 8.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 57 patients will be accrued for this study within 2.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma with expression of bcl-1 and CD20

  * Stage II-IV disease
* Measurable or evaluable disease

  * Measurable disease defined as at least 1 bidimensionally measurable lesion at least 2 cm by imaging scan
  * A spleen at least 17 cm or having discrete filling defects by CT scan will constitute evaluable disease provided that no explanation other than lymphomatous involvement (e.g., portal hypertension or other liver disease) is likely
* No known CNS lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* WBC greater than 2,500/mm^3*
* Platelet count greater than 100,000/mm^3* NOTE: *Unless due to disease in bone marrow

Hepatic

* Bilirubin less than 1.5 mg/dL (1.5-3.0 mg/dL if due to liver involvement by lymphoma)
* ALT and AST no greater than 2.5 times upper limit of normal (unless due to liver involvement by lymphoma)

Renal

* Creatinine less than 2.0 mg/dL
* Calcium no greater than 11.5 mg/dL

Cardiovascular

* LVEF greater than 45%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study participation
* HIV negative
* No other malignancy except treated carcinoma in situ of the cervix or squamous cell or basal cell skin cancer or any other surgically cured malignancy from which the patient has been disease-free for at least 3 years
* No other concurrent serious medical condition or active infection that would preclude ability to deliver standard prednisone, cyclophosphamide, doxorubicin, and vincristine (CHOP) chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior corticosteroids allowed provided the course was no more than 2 weeks in duration

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Smith, MD, PhD, Study Chair — Fox Chase Cancer Center; Leo I. Gordon, MD — Robert H. Lurie Cancer Center
Locations (87):
- United States (81):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Burgess Health Center, Onawa, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (3):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
  - San Juan City Hospital, San Juan
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Smith MR, Zhang L, Gordon LI, et al.: Phase II study of R-CHOP followed by 90Y-ibritumomab tiuxetan in untreated mantle cell lymphoma: Eastern Cooperative Oncology Group study E1499. [Abstract] Blood 110 (11): A-389, 2007.
- [Result] Smith MR, Chen H, Gordon L, et al.: Phase II study of rituximab + CHOP followed by 90Y-ibritumomab tiuxetan in patients with previously untreated mantle cell lymphoma: an Eastern Cooperative Oncology Group Study (E1499). [Abstract] J Clin Oncol 24 (Suppl 18): A-7503, 422s, 2006.